CLINICAL TRIAL: NCT00082758
Title: A Phase II Study Of hu14.18-IL2 In Children With Recurrent Or Refractory Neuroblastoma
Brief Title: hu14.18-Interleukin-2 Fusion Protein in Treating Young Patients With Recurrent or Refractory Neuroblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ANBL0322; CDR0000360723 (Other: Clinical Trials.gov); COG-ANBL0322 (Other: Children's Oncology Group); NCI-2012-02583 (Other: NCI)
Record Dates: First submitted 2004-05-14; First posted 2004-05-19 (Estimated); Results first posted 2014-01-16 (Estimated); Last update posted 2015-02-12 (Estimated); Status verified 2015-01

CONDITIONS: Neuroblastoma
Keywords: recurrent neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — lorukafusp alfa

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Disease Measurable by Standard Criteria(hu14.18-interleukin-2) (Experimental): Patients with residual/refractory neuroblastoma and readily measurable residual/refractory disease using standard radiographic criteria. Standard radiographic criteria for CT/MRI Lesions will use the definitions of measurable disease from the Response Evaluation Criteria In Solid Tumors (RECIST) from the National Cancer Institute.
  hu14.18-Interleukin-2 fusion protein : Given IV
  Interventions: Biological: hu14.18-Interleukin-2 fusion protein
- Disease Eval by MIBG or BM Histology (hu14.18-interleukin-2) (Experimental): Patients with residual/refractory neuroblastoma with disease that is not measurable by standard radiographic criteria, but is evaluable by meta-iodobenzylguanidine (MIBG) scanning and/or by bone marrow (BM) histology.
  hu14.18-Interleukin-2 fusion protein : Given IV
  Interventions: Biological: hu14.18-Interleukin-2 fusion protein
- Disease Identified by BM Immunohistochemistry Only (Experimental): Patients with residual/refractory neuroblastoma that do not have disease that is measurable by standard radiographic techniques or evaluable by meta-iodobenzylguanidine (MIBG) scanning or bone marrow (BM) histology, however, disease is identified and quantified by BM immunohistochemistry (>5 neuroblastoma cells per 1,000,000 nucleated marrow cells).
  hu14.18-Interleukin-2 fusion protein : Given IV
  Interventions: Biological: hu14.18-Interleukin-2 fusion protein

INTERVENTIONS:
Biological: hu14.18-Interleukin-2 fusion protein — Given IV
  Other Names: IMMUNOCYTOKINE HU14.18-IL2 FUSION PROTEIN; humanized anti GD2 antibody fused with human IL-2; BB-IND-9798

SUMMARY:
RATIONALE: Biological therapies such as hu14.18-interleukin-2 fusion protein work in different ways to stimulate the immune system and stop tumor cells from growing.

PURPOSE: This phase II trial is studying how well hu14.18-interleukin-2 fusion protein works in treating young patients with recurrent or refractory neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate in children with recurrent or refractory neuroblastoma treated with hu14.18-interleukin-2 (hu14.18-IL2) fusion protein.
* Determine the adverse events of this drug in these patients.
* Determine the immunologic activation in patients treated with this drug.
* Determine the induction of anti-hu14.18-IL2 antibody in patients treated with this drug.
* Correlate antitumor response with measurements of toxicity, immune activation, and anti-hu14.18-IL2 antibody activity in patients treated with this drug.

OUTLINE: This is a multicenter study. Patients are stratified according to measurable/evaluable disease (measurable by standard radiographic criteria vs evaluable by MIBG (meta-iodobenzylguanidine) scanning and/or bone marrow histology vs disease identified and quantified by bone marrow immunohistochemistry).

For standard radiographic criteria this study will use the definitions of measurable disease from the Response Evaluation Criteria In Solid Tumors (RECIST) from the National Cancer Institute. Complete Response (CR) - Disappearance of all target lesions. No evidence of tumor at any site (chest, abdomen, liver, bone, bone marrow, nodes, etc). Very Good Partial Response (VGPR) - Greater than 90% decrease of the disease measurement for CT/MRI target lesions, taking as reference the disease measurement done to confirm measurable disease in target lesions at study entry; all pre-existing bone lesions with CR by MIBG; MIBG scan can be SD or CR in soft tissue lesions corresponding to lesions on CT/MRI. Partial Response (PR) - At least a 30% decrease in the disease measurement for CT/MRI target lesions, taking as reference the disease measurement done to confirm measurable disease in target lesions at study entry. Progressive Disease (PD) - Any one of the following: a) At least a 20% increase in the disease measurement for CT/MRI target lesions, taking as reference the smallest disease measurement recorded since the start of treatment. b) Appearance of one or more new lesions or new sites of tumor. c) PD as defined above for either bone marrow or MIBG lesions.

Stable disease (SD) - The patient will be classified as stable disease for overall response if there is stable disease by either CT/MRI lesion, bone marrow, or MIBG criteria. No new lesions; no new sites of disease.

Patients will be enrolled in 3 strata, and evaluated for antitumor response following 2 monthly courses (treatment on Days 1-3, followed by 25 days of observation,). Patients with progressive disease will be taken off protocol therapy. Patients with stabilization or regression of disease will be eligible to receive 2 more monthly courses of treatment. Additional treatment following course 4 will be allowed for patients showing a continued clinical response, up to a maximum of 10 courses of treatment.

Patients are followed for survival.

PROJECTED ACCRUAL: A total of 40-60 patients (20 for strata 1 and 2 and 0-20 for stratum 3) will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed neuroblastoma
* Relapsed or refractory to conventional therapy
* Measurable or evaluable disease documented by 1 of the following criteria:

  * Clinical
  * Radiographic
  * Histologic
  * MIBG (meta-iodobenzylguanidine) scanning
  * Immunocytochemistry
* No symptomatic pleural effusions or ascites requiring constant or intermittent drainage
* No clinical or radiological evidence of central nervous system (CNS) disease

PATIENT CHARACTERISTICS:

Age

* 21 and under

Performance status

* Karnofsky 50-100% (> 16 years of age)
* Lansky 50-100% (≤ 16 years of age)

Life expectancy

* At least 8 weeks

Hematopoietic

* Absolute neutrophil count > 1,000/mm^3
* Platelet count ≥ 75,000/mm^3*

  * Must not be refractory to platelet transfusions
* Hemoglobin ≥ 9.0 g/dL* NOTE: *Transfusion allowed if patient is known to have a history of bone marrow involvement with tumor

Hepatic

* Alanine transaminase (ALT) < 2.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* Hepatitis B surface antigen negative

Renal

* Creatinine adjusted according to age as follows:

  * No greater than 0.4 mg/dL (≤ 5 months)
  * No greater than 0.5 mg/dL (6 months -11 months)
  * No greater than 0.6 mg/dL (1 year-23 months)
  * No greater than 0.8 mg/dL (2 years-5 years)
  * No greater than 1.0 mg/dL (6 years-9 years)
  * No greater than 1.2 mg/dL (10 years-12 years)
  * No greater than 1.4 mg/dL (13 years and over [female])
  * No greater than 1.5 mg/dL (13 years to 15 years [male])
  * No greater than 1.7 mg/dL (16 years and over [male]) OR
* Creatinine clearance or radioisotope glomerular filtration rate at least 70 mL/min

Cardiovascular

* Shortening fraction ≥ 27% by echocardiogram OR
* Ejection fraction ≥ 50% by Multi Gated Acquisition Scan (MUGA)
* No symptomatic congestive heart failure
* No uncontrolled cardiac rhythm disturbance

Pulmonary

* Pulse oximetry > 94% on room air
* Forced vital capacity (FVC) > 80%
* Forced expiratory volume (FEV_1) > 80%
* No abnormal respiratory function
* No dyspnea at rest
* No exercise intolerance
* No prior history of ventilator support related to lung injury (e.g., pneumonia, hemorrhagic pneumonitis, or capillary leakage)

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* HIV negative
* No active uncontrolled infection
* No active uncontrolled peptic ulcer
* No objective peripheral neuropathy ≥ grade 2
* No significant psychiatric disabilities
* No seizure disorders requiring antiseizure medications
* No other concurrent significant illness

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Recovered from prior immunotherapy
* Prior in vivo monoclonal antibodies for biologic therapy or tumor imaging allowed provided there is documented absence of detectable antibody to hu14.18 by serology
* More than 28 days since prior autologous stem cell transplantation

  * Prior autologous marrow or stem cell infusion using monoclonal antibody-purged specimens allowed
* More than 1 week since prior growth factors
* At least 7 days since prior nonmyelosuppressive biologic agents
* No prior allogeneic bone marrow or stem cell transplantation
* No concurrent immunomodulating agents
* No concurrent growth factors

Chemotherapy

* More than 3 weeks since prior myelosuppressive chemotherapy (4 weeks for nitrosoureas) and recovered
* No concurrent anticancer chemotherapy

Endocrine therapy

* No concurrent corticosteroids except 100 mg or less of hydrocortisone (or equivalent) as premedication for blood transfusion or treatment for transfusion reaction

  * No other use of systemic steroids

Radiotherapy

* Recovered from prior radiotherapy
* At least 2 weeks since prior local palliative radiotherapy (small port)
* At least 6 months since prior craniospinal radiotherapy
* At least 6 months since prior total body irradiation
* At least 6 months since prior radiotherapy to ≥ 50% of the pelvis
* At least 6 weeks since other prior substantial bone marrow radiotherapy
* Concurrent radiotherapy to localized painful lesions allowed provided at least 1 measurable or evaluable lesion is not irradiated

Surgery

* More than 2 weeks since prior major surgery (e.g., laparotomy or thoracotomy)
* No prior organ allografts

Other

* No concurrent immunosuppressive drugs
* No other concurrent myelosuppressive antineoplastic drugs

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2005-08; Primary Completion 2008-02 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul M Sondel, MD, PhD, Study Chair — University of Wisconsin, Madison; Suzanne Shusterman, MD, Study Chair — Dana-Farber Cancer Institute
Locations (81):
- United States (69):
  - Lurleen Wallace Comprehensive Cancer at University of Alabama - Birmingham, Birmingham, Alabama
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital of Orange County, Orange, California
  - Sutter Cancer Center, Sacramento, California
  - UCSF Comprehensive Cancer Center, San Francisco, California
  - Stanford Comprehensive Cancer Center - Stanford, Stanford, California
  - Children's Hospital Cancer Center, Denver, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - MBCCOP - Medical College of Georgia Cancer Center, Augusta, Georgia
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Markey Cancer Center at University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - Tulane Cancer Center Office of Clinical Research, Alexandria, Louisiana
  - CancerCare of Maine at Eastern Maine Medial Center, Bangor, Maine
  - Floating Hospital for Children at Tufts - New England Medical Center, Boston, Massachusetts
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Spectrum Health Hospital - Butterworth Campus, Grand Rapids, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - University of Minnesota Cancer Center at University of Minnesota, Minneapolis, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Siteman Cancer Center at Barnes-Jewish Hospital, St Louis, Missouri
  - Sunrise Hospital and Medical Center, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth - Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Overlook Hospital, Morristown, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - University of New Mexico Cancer Research and Treatment Center, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - New York Medical College, Valhalla, New York
  - Lineberger Comprehensive Cancer Center at University of North Carolina - Chapel Hill, Chapel Hill, North Carolina
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Columbus Children's Hospital, Columbus, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Geisinger Medical Center, Danville, Pennsylvania
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Palmetto Health South Carolina Cancer Center, Columbia, South Carolina
  - T.C. Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine - Amarillo, Amarillo, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Virginia Commonwealth University Massey Cancer Center, Richmond, Virginia
  - Carilion Cancer Center of Western Virginia, Roanoke, Virginia
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
  - Midwest Children's Cancer Center, Milwaukee, Wisconsin
- Canada (12):
  - Alberta Children's Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Children's & Women's Hospital of British Columbia, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Children's Hospital of Western Ontario, London, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Montreal Children's Hospital at McGill University Health Center, Montreal, Quebec
  - Hopital Sainte Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec

REFERENCES:
- [Result] Delgado DC, Hank JA, Kolesar J, Lorentzen D, Gan J, Seo S, Kim K, Shusterman S, Gillies SD, Reisfeld RA, Yang R, Gadbaw B, DeSantes KB, London WB, Seeger RC, Maris JM, Sondel PM. Genotypes of NK cell KIR receptors, their ligands, and Fcgamma receptors in the response of neuroblastoma patients to Hu14.18-IL2 immunotherapy. Cancer Res. 2010 Dec 1;70(23):9554-61. doi: 10.1158/0008-5472.CAN-10-2211. Epub 2010 Oct 8. PMID 20935224
- [Result] Shusterman S, London WB, Gillies SD, Hank JA, Voss SD, Seeger RC, Reynolds CP, Kimball J, Albertini MR, Wagner B, Gan J, Eickhoff J, DeSantes KB, Cohn SL, Hecht T, Gadbaw B, Reisfeld RA, Maris JM, Sondel PM. Antitumor activity of hu14.18-IL2 in patients with relapsed/refractory neuroblastoma: a Children's Oncology Group (COG) phase II study. J Clin Oncol. 2010 Nov 20;28(33):4969-75. doi: 10.1200/JCO.2009.27.8861. Epub 2010 Oct 4. PMID 20921469

RESULTS

PARTICIPANT FLOW:
Groups:
- Disease Identified by BM Immunohistochemistry Only: Patients with residual/refractory neuroblastoma that do not have disease that is measurable by standard radiographic techniques or evaluable by meta-iodobenzylguanidine (MIBG) scanning or bone marrow (BM) histology, however, disease is identified and quantified by BM immunohistochemistry (>5 neuroblastoma cells per 1,000,000 nucleated marrow cells)
  hu14.18-Interleukin-2 fusion protein : Given IV
Period: Overall Study
Arm/Group | Disease Measurable by Standard Criteria(hu14.18-interleukin-2) | Disease Eval by MIBG or BM Histology (hu14.18-interleukin-2) | Disease Identified by BM Immunohistochemistry Only
Started | 15 | 24 | 0
Completed | 0 | 7 | 0
Not Completed | 15 | 17 | 0
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Lack of Efficacy | 12 | 13 | 0
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Disease Eval by MIBG or BM Histology (hu14.18-interleukin-2): Patients with residual/refractory neuroblastoma with disease that is not measurable by standard radiographic criteria, but is evaluable by MIBG (iodine-131-meta-iodobenzylguanidine) scanning and/or by bone marrow histology.
  hu14.18-Interleukin-2 fusion protein : Given IV
- Disease Identified by BM Immunohistochemistry Only: Patients with residual/refractory neuroblastoma that do not have disease that is measurable by standard radiographic techniques or evaluable by MIBG (iodine-131-meta-iodobenzylguanidine) scanning or BM histology, however, disease is identified and quantified by BM immunohistochemistry (>5 neuroblastoma cells per 1,000,000 nucleated marrow cells).
  hu14.18-Interleukin-2 fusion protein : Given IV
- Total: Total of all reporting groups
Arm/Group | Disease Measurable by Standard Criteria(hu14.18-interleukin-2) | Disease Eval by MIBG or BM Histology (hu14.18-interleukin-2) | Disease Identified by BM Immunohistochemistry Only | Total
Number analyzed (Participants) | 15 | 24 | 0 | 39
Age, Categorical [Number; unit: participants]
  <=18 years | 15 | 23 |  | 38
  Between 18 and 65 years | 0 | 1 |  | 1
  >=65 years | 0 | 0 |  | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 5.98 [4.74 to 10.89] | 6.28 [5.32 to 9.09] |  | 6.16 [4.78 to 9.40]
Gender [Number; unit: participants]
  Female | 7 | 10 |  | 17
  Male | 8 | 14 |  | 22
Ethnicity (NIH/OMB) [Number; unit: participants]
  Hispanic or Latino | 0 | 2 |  | 2
  Not Hispanic or Latino | 15 | 21 |  | 36
  Unknown or Not Reported | 0 | 1 |  | 1
Race (NIH/OMB) [Number; unit: participants]
  American Indian or Alaska Native | 0 | 1 |  | 1
  Asian | 0 | 1 |  | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  | 0
  Black or African American | 5 | 3 |  | 8
  White | 9 | 18 |  | 27
  More than one race | 0 | 0 |  | 0
  Unknown or Not Reported | 1 | 1 |  | 2
Region of Enrollment [Number; unit: participants]
  United States | 14 | 22 |  | 36
  Canada | 1 | 2 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Responders (Response Rate)
Description: Response rate to hu14.18-Interleukin-2 in 3 separate strata of patients with recurrent or refractory neuroblastoma. Patients will have radiologic (CT/MRI) tumor and urine homovanillic acid (HVA)/vanillylmandelic acid (VMA) measurements. Patients with prior marrow involvement will have marrow assessments. Patients with MIBG+ (iodine-131-meta-iodobenzylguanidine) prior disease will have MIBG scans performed. For CT/MRI lesions, measureable disease is measured by the Response Evaluation Criteria In Solid Tumors (RECIST) from the National Cancer Institute. RECIST (v1.0) for target lesions: Complete Response (CR): Disappearance of all target lesions, Partial Response (PR): At least a 30% decrease in the sum of the longest diameter (LD) of target lesions, Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, Progressive Disease (PD): At least a 20% increase in the sum of the LD of target lesions.
Time Frame: Up to 30 weeks
Population: Patients were evaluable for inclusion in the analysis of response if eligible, had an event (relapse, PD, death or secondary malignancy) any time after enrollment, or completed at least 2 courses of Irinotecan/Temozolomide therapy. Patients off therapy before completion of 2 courses by choice or toxicity were not evaluable for response analysis.
Measure: Number; unit: participants
Groups:
- Disease Eval by MIBG or BM Histology (hu14.18-interleukin-2): Patients with residual/refractory neuroblastoma with disease that is not measurable by standard radiographic criteria, but is evaluable by MIBG (meta-iodobenzylguanidine) scanning and/or by bone marrow histology.
  hu14.18-Interleukin-2 fusion protein : Given IV
- Disease Identified by BM Immunohistochemistry Only: Patients with residual/refractory neuroblastoma that do not have disease that is measurable by standard radiographic techniques or evaluable by MIBG (iodine-131-meta-iodobenzylguanidine) scanning or BM histology, however, disease is identified and quantified by BM immunohistochemistry (>5 neuroblastoma cells per 1,000,000 nucleated marrow cells)
  hu14.18-Interleukin-2 fusion protein : Given IV
Arm/Group | Disease Measurable by Standard Criteria(hu14.18-interleukin-2) | Disease Eval by MIBG or BM Histology (hu14.18-interleukin-2) | Disease Identified by BM Immunohistochemistry Only
Number analyzed (Participants) | 13 | 23 | 0
participants
  Responder | 0 | 5 |
  Non-responder | 13 | 18 |

ADVERSE EVENTS:
Time Frame: Duration of protocol therapy
Description: Patients were evaluable for inclusion if they received at least one dose of protocol therapy. SAE field contains NCI Common Terminology Criteria for Adverse Events (CTCAE) submitted via expedited reporting (NCI AdEERs / CAeRs). The AE field contains grade 3 and higher CTCAEs reported on study excluding those that were reported as SAEs.
Arm/Group | Disease Measurable by Standard Criteria(hu14.18-interleukin-2) | Disease Eval by MIBG or BM Histology (hu14.18-interleukin-2) | Disease Identified by BM Immunohistochemistry Only
Serious Adverse Events (participants affected / at risk) | 13/15 | 21/24 | 0/0
Other Adverse Events (participants affected / at risk) | 13/15 | 18/24 | 0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Disease Measurable by Standard Criteria(hu14.18-interleukin-2) (N=15) | Disease Eval by MIBG or BM Histology (hu14.18-interleukin-2) (N=24) | Disease Identified by BM Immunohistochemistry Only (N=0)
Anemia (Blood and lymphatic system disorders) | 3 (4) | 6 (10) | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0
Death NOS (General disorders) | 1 (1) | 0 (0) | 0
Anaphylaxis (Immune system disorders) | 1 (1) | 3 (4) | 0
Bone infection (Infections and infestations) | 0 (0) | 1 (1) | 0
Catheter related infection (Infections and infestations) | 1 (1) | 4 (9) | 0
Infections and infestations (Infections and infestations) | 1 (1) | 0 (0) | 0
Lung infection (Infections and infestations) | 0 (0) | 1 (1) | 0
Tooth infection (Infections and infestations) | 0 (0) | 1 (1) | 0
Alanine aminotransferase (Investigations) | 4 (5) | 4 (6) | 0
Aspartate aminotransferase (Investigations) | 4 (5) | 5 (7) | 0
Blood bilirubin increased (Investigations) | 2 (3) | 6 (8) | 0
GGT increased (Investigations) | 0 (0) | 1 (1) | 0
Lymphocyte count decrease (Investigations) | 4 (8) | 11 (33) | 0
Neutrophil count decreased (Investigations) | 5 (5) | 8 (20) | 0
Platelet count decreased (Investigations) | 5 (6) | 11 (27) | 0
White blood cell decrease (Investigations) | 2 (3) | 7 (12) | 0
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 3 (4) | 0
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Disease Measurable by Standard Criteria(hu14.18-interleukin-2) | Disease Eval by MIBG or BM Histology (hu14.18-interleukin-2) | Disease Identified by BM Immunohistochemistry Only
Anemia (Blood and lymphatic system disorders) | 11/15 (23) | 14/24 (42) | 0/0
Cardiac disorders - Other (Cardiac disorders) | 0/15 (0) | 2/24 (2) | 0/0
Sinus tachycardia (Cardiac disorders) | 1/15 (1) | 7/24 (16) | 0/0
Middle ear inflammation (Ear and labyrinth disorders) | 1/15 (1) | 0/24 (0) | 0/0
Abdominal pain (Gastrointestinal disorders) | 2/15 (2) | 0/24 (0) | 0/0
Ascites (Gastrointestinal disorders) | 2/15 (2) | 0/24 (0) | 0/0
Constipation (Gastrointestinal disorders) | 0/15 (0) | 3/24 (4) | 0/0
Diarrhea (Gastrointestinal disorders) | 1/15 (2) | 6/24 (10) | 0/0
Nausea (Gastrointestinal disorders) | 2/15 (2) | 0/24 (0) | 0/0
Vomiting (Gastrointestinal disorders) | 2/15 (3) | 8/24 (18) | 0/0
Chills (General disorders) | 1/15 (1) | 0/24 (0) | 0/0
Edema face (General disorders) | 3/15 (3) | 9/24 (17) | 0/0
Edema limbs (General disorders) | 3/15 (5) | 2/24 (5) | 0/0
Edema trunk (General disorders) | 1/15 (1) | 3/24 (4) | 0/0
Fever (General disorders) | 1/15 (1) | 0/24 (0) | 0/0
Localized edema (General disorders) | 1/15 (1) | 0/24 (0) | 0/0
Otitis media (Infections and infestations) | 0/15 (0) | 2/24 (2) | 0/0
Pharyngitis (Infections and infestations) | 0/15 (0) | 2/24 (2) | 0/0
Sinusitis (Infections and infestations) | 1/15 (1) | 0/24 (0) | 0/0
Upper respiratory infection (Infections and infestations) | 1/15 (1) | 0/24 (0) | 0/0
Bruising (Injury, poisoning and procedural complications) | 1/15 (1) | 0/24 (0) | 0/0
Alanine aminotransferase (Investigations) | 10/15 (20) | 14/24 (41) | 0/0
Alkaline phosphatase increased (Investigations) | 2/15 (2) | 5/24 (7) | 0/0
Aspartate aminotransferase (Investigations) | 9/15 (17) | 15/24 (44) | 0/0
Blood bilirubin increased (Investigations) | 9/15 (13) | 9/24 (22) | 0/0
Cholesterol high (Investigations) | 1/15 (2) | 0/24 (0) | 0/0
Creatinine increased (Investigations) | 3/15 (6) | 4/24 (6) | 0/0
GGT increased (Investigations) | 1/15 (2) | 4/24 (9) | 0/0
Investigations - Other (Investigations) | 0/15 (0) | 2/24 (26) | 0/0
Lymphocyte count decrease (Investigations) | 1/15 (1) | 4/24 (8) | 0/0
Neutrophil count decreased (Investigations) | 5/15 (6) | 6/24 (14) | 0/0
Platelet count decreased (Investigations) | 8/15 (17) | 11/24 (22) | 0/0
Weight gain (Investigations) | 3/15 (3) | 6/24 (12) | 0/0
White blood cell decrease (Investigations) | 9/15 (16) | 10/24 (32) | 0/0
Acidosis (Metabolism and nutrition disorders) | 2/15 (2) | 3/24 (4) | 0/0
Anorexia (Metabolism and nutrition disorders) | 4/15 (4) | 3/24 (8) | 0/0
Dehydration (Metabolism and nutrition disorders) | 1/15 (1) | 0/24 (0) | 0/0
Hypercalcemia (Metabolism and nutrition disorders) | 1/15 (1) | 0/24 (0) | 0/0
Hyperglycemia (Metabolism and nutrition disorders) | 7/15 (13) | 13/24 (26) | 0/0
Hyperkalemia (Metabolism and nutrition disorders) | 1/15 (1) | 2/24 (2) | 0/0
Hypermagnesemia (Metabolism and nutrition disorders) | 0/15 (0) | 3/24 (4) | 0/0
Hypernatremia (Metabolism and nutrition disorders) | 1/15 (1) | 2/24 (2) | 0/0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1/15 (2) | 0/24 (0) | 0/0
Hypoalbuminemia (Metabolism and nutrition disorders) | 10/15 (20) | 15/24 (45) | 0/0
Hypocalcemia (Metabolism and nutrition disorders) | 8/15 (17) | 14/24 (38) | 0/0
Hypoglycemia (Metabolism and nutrition disorders) | 0/15 (0) | 3/24 (8) | 0/0
Hypokalemia (Metabolism and nutrition disorders) | 4/15 (5) | 7/24 (17) | 0/0
Hypomagnesemia (Metabolism and nutrition disorders) | 6/15 (14) | 8/24 (13) | 0/0
Hyponatremia (Metabolism and nutrition disorders) | 4/15 (11) | 11/24 (27) | 0/0
Hypophosphatemia (Metabolism and nutrition disorders) | 8/15 (14) | 11/24 (20) | 0/0
Bone pain (Musculoskeletal and connective tissue disorders) | 1/15 (1) | 0/24 (0) | 0/0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1/15 (1) | 0/24 (0) | 0/0
Intracranial hemorrhage (Nervous system disorders) | 1/15 (1) | 0/24 (0) | 0/0
Anxiety (Psychiatric disorders) | 0/15 (0) | 2/24 (3) | 0/0
Renal and urinary disorders, Other (Renal and urinary disorders) | 0/15 (0) | 3/24 (3) | 0/0
Urinary retention (Renal and urinary disorders) | 1/15 (1) | 0/24 (0) | 0/0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0/15 (0) | 2/24 (2) | 0/0
Cough (Respiratory, thoracic and mediastinal disorders) | 4/15 (5) | 3/24 (7) | 0/0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1/15 (1) | 2/24 (3) | 0/0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1/15 (1) | 5/24 (5) | 0/0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0/15 (0) | 2/24 (2) | 0/0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1/15 (1) | 3/24 (5) | 0/0
Respiratory, thoracic and mediastinal disorders, Other (Respiratory, thoracic and mediastinal disorders) | 0/15 (0) | 2/24 (3) | 0/0
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1/15 (1) | 0/24 (0) | 0/0
Alopecia (Skin and subcutaneous tissue disorders) | 0/15 (0) | 2/24 (2) | 0/0
Dry skin (Skin and subcutaneous tissue disorders) | 1/15 (1) | 5/24 (12) | 0/0
Pruritus (Skin and subcutaneous tissue disorders) | 2/15 (4) | 6/24 (10) | 0/0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1/15 (1) | 0/24 (0) | 0/0
Flushing (Vascular disorders) | 0/15 (0) | 2/24 (2) | 0/0
Hypertension (Vascular disorders) | 1/15 (1) | 3/24 (3) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.